CLINICAL TRIAL: NCT06557668
Title: Clinical Outcomes of Treatment With Immunomodulator Plus Standard Anti-cancer Therapies for Patients With Colorectal Cancer: A Retrospective Study
Brief Title: Clinical Outcomes of Treatment With Immunomodulator Plus Cancer Therapies for Patients With Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Chou-Chen Chen, Attending Physician, Taichung Veterans General Hospital
Other Study IDs: APS-CRC01
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Astragalus Polysaccharides; Survival
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer treatment with immunomodulator: CRC patients had previously received cancer therapies along with immunomodulator
- Cancer treatment without immunomodulator: CRC patients had previously received cancer therapies without immunomodulator

SUMMARY:
This study aims to evaluate the survival and treatment outcomes among colorectal cancer patients undergoing anti-cancer treatment, both with and without an immunomodulator.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide. The clinical outcomes from CRC treatments are often unsatisfactory for the majority of patients. The tumor microenvironment (TME) plays an important role to regulate tumor growth, progression, and metastasis and can limit the efficacy of cancer therapies. Therefore, targeting TME could provide an efficient approach for cancer treatment.

Astragalus Polysaccharide Injection, an immunomodulator, which can stimulate medullary hematopoiesis and enhance immune function. It also can modulate TME. Astragalus Polysaccharide Injection has been approved as a prescription drug for alleviating cancer-related fatigue by the Taiwan Food and Drug Administration (TFDA).

In this retrospective study, we will collect clinical data and survival status of colorectal cancer patients undergoing anti-cancer treatment from their medical records with and without immunomodulator, Astragalus polysaccharide Injection. It can be used to understand the possible clinical benefit of immunomodulator plus anti-cancer therapies for patients with colorectal cancer, and physicians can refer to these results to give patients the suitable treatment recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years and older.
* Patients who have been given a diagnosis of colorectal cancer.
* Patients had previously initiated anti-cancer therapies between January 1, 2020, and Apr 30, 2024.

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal Cancer
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the initial treatment until April 2024

SECONDARY OUTCOMES:
Progress free survival | From the initial treatment until April 2024
Tumor response | From the initial treatment until April 2024

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chung-Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung

IPD SHARING:
Plan to Share IPD: Undecided